CLINICAL TRIAL: NCT07033715
Title: Effects of a 12-week Exercise Intervention on Physical and Mental Health in Hereditary ATTR (ATTRv) Amyloidosis
Brief Title: Exercise in Hereditary ATTR (ATTRv) Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Cláudia Barata, Principal Investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 212/2024; 2023.00324.BD (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2025-04-18; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Amyloidosis, Hereditary, Transthyretin-Related
Keywords: ATTRv; exercise; physical fitness; mental health; HRQoL
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will be enrolled in a 12-week supervised exercise intervention.
  Interventions: Other: Exercise
- Control (No Intervention): Participants will not be enrolled in the 12-week exercise program.

INTERVENTIONS:
Other: Exercise — The exercise sessions will have a frequency of 3 times a week and a duration of 60 minutes per session. Exercise intensity will be gradually increased throughout the program and will be monitored every session using Borg's Rated Perceived Exertion scale, aiming at levels of 12-13 ("fairly light to somewhat hard"). The program will be mainly composed of cardiorespiratory exercises and resistance exercises. It will also comprise flexibility exercises to improve joint range of motion and neuromotor exercises involving motor skills (balance, agility, coordination, gait...), proprioceptive training and multifaceted activities (tai ji, yoga...).
  Arms: Exercise

SUMMARY:
This study aims to explore the effects of a 12-week exercise intervention on the physical and mental health of people living with Hereditary ATTR (ATTRv) Amyloidosis, a rare genetic disease caused by mutations in the transthyretin gene, leading to the deposition of amyloid fibrils in nerves and organs.

DETAILED DESCRIPTION:
Considering that few studies to date have explored the effects of exercise in ATTRv Amyloidosis, this study aims to increase the existing evidence in this under-researched area. Besides, the existing research was performed with liver transplanted patients and focused exclusively on physical fitness outcomes. Therefore, we aim to include those patients who are currently receiving new therapies and extend research to the mental benefits of exercising, questioning whether exercise can ease the mental burden of living with such a debilitating disease. This research also seeks to raise awareness among patients and healthcare professionals about the importance of an active lifestyle in improving HRQoL in this community.

ELIGIBILITY:
Inclusion Criteria:

* ATTRv Amyloidosis patients living in Portugal;
* Disease stage 1 or 2;
* No medical contraindication for exercising;
* Ability to provide informed consent.

Exclusion Criteria:

- Having undergone a liver transplant in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Strength of the knee extensors | Strength of the knee extensors will be assessed at baseline and immediately after the 12-week exercise intervention.
  The strength of the knee extensors (N) will be assessed with a handheld strength device (DynaMo, VALD Performance).
Grip strength | Grip strength will be assessed at baseline and immediately after the 12-week exercise intervention.
  Grip strength (N) will be assessed with a handheld strength device (DynaMo, VALD Performance).
Walking capacity | Walking capacity will be assessed at baseline and immediately after the 12-week exercise intervention.
  Walking capacity will be assessed with the 6-minute walk test, registering the total distance covered in the test (m).
Body mass index | Body mass index will be assessed at baseline and immediately after the 12-week exercise intervention.
  Body mass index (kg/m^2) will be calculated from the ratio between weight and the square of height.
Weight | Weight will be assessed at baseline and immediatly after the 12-week exercise intervention.
  Weight (kg) will be assessed with a bioelectrical impedance device (TANITA BC-545N).
Fat free mass | Fat free mass will be assessed at baseline and immediately after the 12-week exercise intervention.
  Fat free mass (kg) will be assessed with a bioelectrical impedance device (TANITA BC-545N).
Fat mass | Fat mass will be assessed at baseline and immediately after the 12-week exercise intervention.
  Fat mass (%) will be assessed with a bioelectrical impedance device (TANITA BC-545N).
Body water | Body water will be assessed at baseline and immediately after the 12-week exercise intervention.
  Body water (kg) will be assessed with a bioelectrical impedance device (TANITA BC-545N).

SECONDARY OUTCOMES:
Mental health | Mental health will be assessed at baseline and immediately after the 12-week exercise intervention.
  Mental health will be evaluated using the Portuguese adaptation of the Mental Health Continuum-Short Form (MHC-SF), a mental-health questionnaire with 14 items that investigates respondent's emotional (3 items), social (5 items) and psychological (6 items) well-being. Each item is rated on a 6-point Likert scale, ranging from 0 (never) to 5 (everyday).

OTHER OUTCOMES:
Health-related quality of life (HRQoL) | HRQoL will be assessed at baseline and immediately after the 12-week exercise intervention.
  To assess HRQoL, the EQ-5D-3L will be used to determine patients' health state in 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2) and extreme problems (3).

CONTACTS AND LOCATIONS:
Overall Officials: João L. Viana, PhD, Study Director — University of Maia
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
The study will involve the collection of sensitive personal data regarding patient's physical and mental health.